CLINICAL TRIAL: NCT06091137
Title: Altered Gut Microbiome Composition by Appendectomy Contributes to Colorectal Cancer
Brief Title: Appendectomy and Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jun YU, Professor, Chinese University of Hong Kong
Other Study IDs: 2022.203
Record Dates: First submitted 2023-10-08; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer; Appendicitis
MeSH Terms: conditions — Colorectal Neoplasms; Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-appendectomy controls
- Appendectomy cases

SUMMARY:
Colorectal cancer (CRC) is one of the most common cancer worldwide. Initiation and progression of CRC involve complex interactions among genetic, epigenetic and environmental factors. Given that hereditary and familial CRC only accounts for 2% to 5% of cases, environmental factors are the key triggers of CRC. Emerging evidence has indicated that gut microbes are an important environmental factor promoting CRC development. Gut dysbiosis has been shown to promote colorectal carcinogenesis in mice. Several individual bacterial species, such as the enterotoxigenic Bacteroides fragilis (ETBF), Fusobacterium nucleatum and Peptostreptococcus anaerobius, could exert carcinogenic effects by inducing direct DNA damage, oxidative damage and activating oncogenic signaling pathways. Recent studies have shown that the appendix plays an important role in maintaining homeostasis and biodiversity of gut microbiome by providing an ideal ecological niche for commensal bacteria and production of immunoglobulin A. Considering the key role of microorganisms in gastrointestinal pathophysiology, absence of appendix may result in disruption of microbiome homeostasis, which could potentially influence the risk of developing CRC. In terms of epidemiological evidence, the association of appendectomy with the risk of CRC development has been controversial, and to date no consensus has been attained. Although gut microorganisms could be a crucial pivot between appendectomy and risk of subsequent CRC development, the direct contribution of appendectomy and the underlying mechanisms are still largely unexplored. In this study, we aim to study

1. the association between appendectomy and colorectal cancer, and
2. the role of appendectomy in CRC risk through causing gut microbial dysbiosis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals underwent appendectomy from January 2000 to December 2020

Exclusion Criteria:

1. patients with the age ≤18 years at enrollment;
2. Patients with any malignant diseases or inflammatory bowel disease history before enrollment;
3. Patients with hereditary syndromes of colorectal adenomas or polyps (familial adenomatous polyposis, Lynch syndrome, etc.);
4. Patients that underwent appendectomy for appendiceal neoplasms.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 60000 appendectomy cases and 120000 controls
Sampling Method: Non-Probability Sample
Enrollment: 180000 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Appendectomy is associated with risk of subsequent CRC incidence | 3 years
  Individuals underwent appendectomy from January 2000 to December 2020 will be retrieved from a population-based database (CDARS) in Hong Kong. For the control group, individuals without appendectomy between 2000 and 2020 based on the same exclusion criteria will be identified from the total population register of CDARS. For each case of appendectomy, we will select two matched referential individuals from the pool based on the year of birth and gender to study the association between appendectomy and CRC risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Digestive Disease, The Chinese University of Hong Kong, Shatin, Hong Kong